CLINICAL TRIAL: NCT05173792
Title: A Phase I, Multicenter, Open-Label, Dose-escalation and Dose-exploration Study to Evaluate the Safety, Pharmacokinetics, and Anti-tumor Activity of of AK119 (CD73) in Subjects With Advanced Solid Tumors
Brief Title: Study of AK119 in Subjects With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AK119-103
Record Dates: First submitted 2021-11-23; First posted 2021-12-30 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Solid Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AK119 (Experimental): Subjects will receive escalating doses of AK119 every 2 or 3 weeks.
  Interventions: Drug: AK119

INTERVENTIONS:
Drug: AK119 — Subjects will receive AK119 intravenously.

SUMMARY:
This is Phase 1, Multicenter, Open-Label, Dose-Escalation and Dose-Exploration Study to Evaluate the Safety, Pharmacokinetics, and Anti-tumor Activity of AK119 (Anti-CD73) in Subjects with Advanced or Metastatic Solid Tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Eastern Cooperative Oncology Group (ECOG) Performance Status 0 to1.
3. Life expectancy ≥12 weeks;
4. Females of childbearing potential must be willing to use a highly effective method of birth control for the duration of the study, and within 120 days after the last dose of investigational product.
5. Non-sterile males must be willing to use a highly effective method of birth control for the duration of the study and within 120 days after the last dose of investigational product.
6. Subjects must have histologically or cytologically confirmed advanced or metastatic solid tumor that is refractory or relapsed to the current standard therapies, or for which no effective standard therapy is available, or whereby standard therapy has been refused.
7. Subjects must have evaluable lesions according to RECIST v1.1.
8. Adequate organ function.

Exclusion Criteria:

1. Prior malignancy active within the previous 3 years except for the tumor for which a subject is enrolled in the study, and locally curable cancers that have been apparently cured.
2. Receipt of the following treatments or procedures:

   1. Anticancer small-molecule targeted agent (e.g., tyrosine kinase inhibitor) within 2 weeks prior to the first dose of investigational product;
   2. Anti-PD-1/PD-L1 mAb within 4 weeks prior to the first dose of investigational product;
   3. Prior use of approved or investigational anti-CTLA-4 therapy, anti-CD73 therapy or adenosine 2A receptor inhibitors, or any other antibody or drug targeting T cell costimulation or immune checkpoint pathways such as ICOS, or agonists such as CD40, CD137, GITR, OX40 etc.;
   4. Other anticancer mAb within 4 weeks or 5 half-lives (whichever is less) prior to the first dose of investigational product;
   5. Other anticancer therapy (e.g., chemotherapy, radiotherapy, etc.) within 4 weeks prior to the first dose of investigational product;
   6. Any major surgery within 4 weeks prior to the first dose of investigational product;
   7. Any other non-approved investigational product or procedure within 4 weeks prior to the first dose of investigational product, or concurrent participation in another therapeutic clinical study;
   8. Any topical therapy (e.g., TACE, HAIC, TARE) within 4 weeks prior to the first dose of investigational product;
3. Subjects with history of brain metastases that have been treated may participate provided they show evidence of stable supra-tentorial lesions at Screening;
4. Brain stem metastasis, meningeal metastasis, spinal cord metasasis or compression;
5. Uncontrolled massive ascites, pleural effusion or pericardial effusion, as determined by the Investigator;
6. Known history of human immunodeficiency virus (HIV) infection;
7. Known active hepatitis B or C infections (Active hepatitis B is defined as a known positive Hepatitis B surface antigen [HBsAg] result. Active hepatitis C is defined by a known positive Hepatitis C virus [HCV] antibody with detectable HCV ribonucleic acid [RNA] results);
8. Active autoimmune diseases or history of autoimmune diseases that may relapse;
9. History of interstitial lung disease, noninfectious pneumonitis except for those induced by radiation therapies;
10. Patients with clinically significant cardio-cerebrovascular or venous thromboembolic disease;
11. Toxicities of prior anticancer therapy have not resolved to NCI-CTCAE version 5.0 Grade ≤1, or to levels dictated in the inclusion/exclusion criteria, except toxicities not considered a safety risk (e.g., alopecia, neuropathy, or asymptomatic laboratory abnormalities);
12. History of severe hypersensitivity reactions to other mAbs;
13. Prior organ transplantation;
14. Any condition that required systemic treatment with corticosteroids (> 10 mg daily prednisone or equivalent) or other immunosuppressive agents within 14 days prior to the first dose of investigational product;
15. Receipt of live attenuated vaccines within 4 weeks prior to the first dose of investigational product; Note: seasonal vaccine for influenza which is generally inactivated is allowed;
16. Any other conditions that, in the opinion of the Investigator, would interfere with evaluation of the investigational product or interpretation of subject safety or study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-12-22 (Actual); Primary Completion 2023-05-22 (Actual); Study Completion 2023-05-22 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) | From the time of informed consent signed through 90 days after the last dose of study drug
  An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product temporally associated with the use of study treatment, whether or not considered related to the study treatment.
Number of participants with a Dose Limiting Toxicity (DLT) | During the first 4 weeks in dose-escalation phase, during the first 3 weeks in dose-exploration phase
  DLTs will be assessed during the first 4 weeks of treatment for dose-escalation phase and first 3 weeks for dose-exploration phase. DLTs are defined as toxicities that meet pre-defined severity criteria, and assessed as having a suspected relationship to study drug, and unrelated to disease, disease progression, inter-current illness, or concomitant medications that occurs within the DLT observation period.

SECONDARY OUTCOMES:
Serum PK concentration of AK119 | From first dose of study drug through 30 days after last dose of study drug
  Serum PK concentration of AK119 in individual subjects at different time points after AK119 administration.
Number of subjects who develop detectable anti-drug antibodies (ADAs) | From first dose of study drug through 90 days after last dose of study drug
  The immunogenicity of AK119 will be assessed by summarizing the number of subjects who develop detectable anti-drug antibodies (ADAs).
Objective response rate (ORR) | Up to 2 years
  ORR is defined as the proportion of subjects with confirmed CR or confirmed PR.
Disease control rate (DCR) | Up to 2 years
  DCR is defined as the proportion of subjects with CR, PR, or SD.
Progression-free survival (PFS) | Up to 2 years
  PFS is defined as the time from the start of treatment with AK119 until the first documentation of disease progression or death due to any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Jihui Hao, PhD, Principal Investigator — Tianjin Medical University Cancer Insitute & Hospital; Tianshu Liu, Principal Investigator — Shanghai Zhongshan Hospital
Locations (2):
- China (2):
  - Fudan University Zhongshan Hospital, Shanghai
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin